CLINICAL TRIAL: NCT01809795
Title: The Health Effects of a Blueberry Enriched Diet on Obese Children: A Feasibility Study
Brief Title: The Health Effects of a Blueberry Enriched Diet on Obese Children
Acronym: Wild Blueberry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Pennington Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-4400
Record Dates: First submitted 2013-02-06; First posted 2013-03-13 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Obesity
Keywords: Obesity; Exercise; Blueberry Plant
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blueberry Smoothie (Experimental): Participants in this group will receive a smoothie containing 1 1/2 cups of freeze-dried whole blueberries crushed into a powder.
  Interventions: Other: Blueberry Smoothie
- Sham Smoothie (Sham Comparator): Participants in this group will receive a smoothie that contains no blueberries.
  Interventions: Other: Sham Smoothie

INTERVENTIONS:
Other: Blueberry Smoothie
  Arms: Blueberry Smoothie
Other: Sham Smoothie
  Arms: Sham Smoothie

SUMMARY:
The purpose of this study to determine if adding blueberries to obese children's diet will improve weight status and other medical testing. We would also like to determine if a larger research study involving blueberries is possible.

DETAILED DESCRIPTION:
Ten children aged 12 to 17 years of age who have a BMI > 95th percentile for age and who are patients of the Center for Better Health and Nutrition will be recruited for this 12 week study.

Group 1 (Standard Therapy): Participants will be asked not to consume berries during the study so as not to confound the effects of eating blueberries. They will, however, be encouraged to consume other fruits consistent with nutrition guidelines for the Healthy Eating Plan (HEP: reduced glycemic load diet).

Participants will be instructed and receive educational handout materials on implementing HEP. In addition participants will be introduced to the use of behavioral tools (e.g. goal setting, daily tracking when goals are met, and incentives provided by the family) to help them stay on track with HEP. Participants will be seen by the dietitian at monthly intervals consistent with programmatic standard of care to review adherence to HEP, use of behavioral tools, and change in weight status.

Participants will be encouraged to attend group exercise classes five days per week or a minimum of four days per week. At the end of each exercise session, participants will receive a "sham smoothie" which contains no blueberries. The children will be directly observed by a study worker when consuming the smoothies to ensure compliance and measure how much of the smoothie was consumed.

Group 2 (Blueberry Enhanced): All the features of Group 1 with the exception that the participants will be given a smoothie that contain 1 1/2 cups of freeze-dried whole blueberries crushed into a powder per serving.

ELIGIBILITY:
Inclusion Criteria:

* Children 12 to 17 years old at the time of enrollment
* Children with a BMI ≥ 95th percentile for age
* Children participating in a weight management program at the CBHN.

Exclusion Criteria:

* Children/parents/guardians who appear unable to understand the study
* Children/parents appear unable to meet the requirements of participating, specifically not missing more than 1 consecutive week during the 12 week intervention
* Children who have a medical condition or development impairment that precludes them from participating in an exercise program
* Children who have type 2 diabetes
* Children who have been diagnosed with hypertension
* Children who are taking a statin
* Children who are pregnant or have given birth within 6 months
* Children with a history of significant cardiac disease leading to cardiovascular instability
* Children who have food allergies or are lactose intolerant
* Children who are unable to finish at least half of the smoothie while they taste it after the consent/assent process or decide after tasting the smoothie that they are no longer interested in participating.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2013-03; Primary Completion 2013-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Attendance and compliance to healthy eating plan, group exercise class and smoothie consumption will be measured to assess feasibility of larger, randomized study. | 12 weeks

SECONDARY OUTCOMES:
Vascular Function | Baseline and after 12 week program
  Vascular Function Testing: augmentation index, Brachial Arterial Distensibility, Pulse Wave Velocity, EndoPAT, Laser Flow Doppler, Ultrasound Brachial Flow Mediated Dilation.
Graded Exercise Test | Baseline and after 12 week program
  Exercise data: graded exercise test with submaximal VO2 measure at 6 and 9 minutes, VO2 max values.
Cognitive Function/Memory | Baseline and after 12 week program
  Cognitive Function/Memory-CVLT and D-KFES at the initial medical evaluation and the WRAMIL 2-D-KFES Alternative Version at the final medical evaluation.
Anthropometric Measurements | Baseline and after 12 week program
  Anthropometrics and clinical measurements: height, weight, BMI, BMI percentile, waist circumference, blood pressure, percent body fat by bioimpedance.
Laboratory Testing | Baseline and after 12 week program
  Laboratory testing: fasting blood sugar, insulin, HDL, LDL, Total Cholesterol, Triglycerides, HgA1C, AST, ALT, GGT for research purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Siegel, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Ogden CL, Carroll MD, Curtin LR, Lamb MM, Flegal KM. Prevalence of high body mass index in US children and adolescents, 2007-2008. JAMA. 2010 Jan 20;303(3):242-9. doi: 10.1001/jama.2009.2012. Epub 2010 Jan 13. PMID 20071470
- [Background] Freedman DS, Khan LK, Serdula MK, Dietz WH, Srinivasan SR, Berenson GS. The relation of childhood BMI to adult adiposity: the Bogalusa Heart Study. Pediatrics. 2005 Jan;115(1):22-7. doi: 10.1542/peds.2004-0220. PMID 15629977
- [Background] Deckelbaum RJ, Williams CL. Childhood obesity: the health issue. Obes Res. 2001 Nov;9 Suppl 4:239S-243S. doi: 10.1038/oby.2001.125. PMID 11707548
- [Background] Lampe JW. Health effects of vegetables and fruit: assessing mechanisms of action in human experimental studies. Am J Clin Nutr. 1999 Sep;70(3 Suppl):475S-490S. doi: 10.1093/ajcn/70.3.475s. PMID 10479220
- [Background] Prior RL. Fruits and vegetables in the prevention of cellular oxidative damage. Am J Clin Nutr. 2003 Sep;78(3 Suppl):570S-578S. doi: 10.1093/ajcn/78.3.570S. PMID 12936951
- [Background] Duffy KB, Spangler EL, Devan BD, Guo Z, Bowker JL, Janas AM, Hagepanos A, Minor RK, DeCabo R, Mouton PR, Shukitt-Hale B, Joseph JA, Ingram DK. A blueberry-enriched diet provides cellular protection against oxidative stress and reduces a kainate-induced learning impairment in rats. Neurobiol Aging. 2008 Nov;29(11):1680-9. doi: 10.1016/j.neurobiolaging.2007.04.002. Epub 2007 May 23. PMID 17524525
- [Background] Wu X, Kang J, Xie C, Burris R, Ferguson ME, Badger TM, Nagarajan S. Dietary blueberries attenuate atherosclerosis in apolipoprotein E-deficient mice by upregulating antioxidant enzyme expression. J Nutr. 2010 Sep;140(9):1628-32. doi: 10.3945/jn.110.123927. Epub 2010 Jul 21. PMID 20660283
- [Background] Wang YP, Cheng ML, Zhang BF, Mu M, Wu J. Effects of blueberry on hepatic fibrosis and transcription factor Nrf2 in rats. World J Gastroenterol. 2010 Jun 7;16(21):2657-63. doi: 10.3748/wjg.v16.i21.2657. PMID 20518088
- [Background] Casadesus G, Shukitt-Hale B, Stellwagen HM, Zhu X, Lee HG, Smith MA, Joseph JA. Modulation of hippocampal plasticity and cognitive behavior by short-term blueberry supplementation in aged rats. Nutr Neurosci. 2004 Oct-Dec;7(5-6):309-16. doi: 10.1080/10284150400020482. PMID 15682927
- [Background] Andres-Lacueva C, Shukitt-Hale B, Galli RL, Jauregui O, Lamuela-Raventos RM, Joseph JA. Anthocyanins in aged blueberry-fed rats are found centrally and may enhance memory. Nutr Neurosci. 2005 Apr;8(2):111-20. doi: 10.1080/10284150500078117. PMID 16053243
- [Background] Elks CM, Reed SD, Mariappan N, Shukitt-Hale B, Joseph JA, Ingram DK, Francis J. A blueberry-enriched diet attenuates nephropathy in a rat model of hypertension via reduction in oxidative stress. PLoS One. 2011;6(9):e24028. doi: 10.1371/journal.pone.0024028. Epub 2011 Sep 15. PMID 21949690
- [Background] Kay CD, Holub BJ. The effect of wild blueberry (Vaccinium angustifolium) consumption on postprandial serum antioxidant status in human subjects. Br J Nutr. 2002 Oct;88(4):389-98. doi: 10.1079/BJN2002665. PMID 12323088
- [Background] Stull AJ, Cash KC, Johnson WD, Champagne CM, Cefalu WT. Bioactives in blueberries improve insulin sensitivity in obese, insulin-resistant men and women. J Nutr. 2010 Oct;140(10):1764-8. doi: 10.3945/jn.110.125336. Epub 2010 Aug 19. PMID 20724487
- [Background] Krikorian R, Shidler MD, Nash TA, Kalt W, Vinqvist-Tymchuk MR, Shukitt-Hale B, Joseph JA. Blueberry supplementation improves memory in older adults. J Agric Food Chem. 2010 Apr 14;58(7):3996-4000. doi: 10.1021/jf9029332. PMID 20047325
- [Background] Basu A, Du M, Leyva MJ, Sanchez K, Betts NM, Wu M, Aston CE, Lyons TJ. Blueberries decrease cardiovascular risk factors in obese men and women with metabolic syndrome. J Nutr. 2010 Sep;140(9):1582-7. doi: 10.3945/jn.110.124701. Epub 2010 Jul 21. PMID 20660279
- [Background] Barlow SE; Expert Committee. Expert committee recommendations regarding the prevention, assessment, and treatment of child and adolescent overweight and obesity: summary report. Pediatrics. 2007 Dec;120 Suppl 4:S164-92. doi: 10.1542/peds.2007-2329C. PMID 18055651
- [Background] Kirk S, Brehm B, Saelens BE, Woo JG, Kissel E, D'Alessio D, Bolling C, Daniels SR. Role of carbohydrate modification in weight management among obese children: a randomized clinical trial. J Pediatr. 2012 Aug;161(2):320-7.e1. doi: 10.1016/j.jpeds.2012.01.041. Epub 2012 Feb 28. PMID 22381024